CLINICAL TRIAL: NCT00809796
Title: A Phase I/II Clinical Study Using Pentamidine in Patients With Metastatic Colon Cancer Undergoing Standard Folinic Acid, 5-Fluorouracil, or Capecitabine and Oxaliplatin Chemotherapy as Second-line and/or Third-line Treatment
Brief Title: A Safety Study of Pentamidine in Patients With Metastatic Colon Cancer Undergoing Standard Chemotherapy as Second-line and/or Third-line Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncozyme Pharma Inc. (Industry)
Responsible Party: Dr. Terry Chow/President, Oncozyme Pharma Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-103
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Use of pentamidine in second and/or third line metastatic colon cancer
  Interventions: Drug: pentamidine

INTERVENTIONS:
Drug: pentamidine — one dose of 4 mg/kg to two dose of 4 mg/kg with possibility of escalated to two dose of 6 mg/kg with or without standard chemotherapy.

SUMMARY:
The purpose of this study is to investigate the safety and possible efficacy of the use of pentamidine in the treatment of colon cancer metastasis in subjects receiving standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of adenocarcinoma of the colon or rectum with evidence of (1) unresectable, locally recurrent, or (2) metastatic disease
* Failure of first-line or second-line therapy for colorectal cancer
* At least one unidimensional measurable lesion (on spiral CT scan)
* 18 years of age or older
* ECOG performance status 0, 1 or 2
* Serum aspartate transaminase (AST) serum alanine transaminase (ALT) £ 2.5 x upper limit of normal (ULN), or AST and ALT £ 5 x ULN if liver function abnormalities are due to underlying malignancy
* Total serum bilirubin £ 1.5 x ULN
* Serum albumin ≥ 3.0 g/dL
* lipase within normal limits
* Absolute neutrophil count (ANC) ≥ 1500/uL (1.5 x 109/L)
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine £ 1.5 x ULN or calculated creatinine clearance ≥ 50 ml/min
* Magnesium ≥ lower limit of normal
* CEA level ≥ 3.4 ng/ml
* Normal ECG
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures
* Life expectancy, in the opinion of the investigator, > 3 months

Exclusion Criteria:

* BP < 100 (systolic)
* History of renal disease, pancreatitis, or diabetes mellitus
* Peripheral sensory neuropathy (> Grade 1, as per NCI CTCAE version 3.0)
* Concomitant therapy with other investigational agents or participation in another clinical trial
* Any of the following conditions: Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2; atrial fibrillation of any grade; QTc interval >450 msec for males or >470 msec for females or uncontrolled intercurrent illness, e.g., unstable angina; severe coronary disease, ventricular arrhythmias, bradycardia <50 bpm
* Active uncontrolled bacterial infection
* Concurrent use of drugs that could prolong QT interval
* Concurrent use of nephrotoxic drugs, including aminoglycosides, ampho B, foscarnet, cidofovir
* Concurrent use of drugs that may be associated with pancreatitis
* Concurrent active cancer originating from a primary site other than colon/rectum, except for surgically treated nonmelanoma skin cancer, in situ cervical cancer, or localized prostate cancer with undetectable PSA level
* Co-existing lung disease
* History of allergy or hypersensitivity to pentamidine Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to first dose of study medication.
* Severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with trial participation of study drug administration, or which in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* On oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Any severe events, tumor marker CEA, and tumor size (CT scan) | Three Months

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kavan, MD, Ph.D., Principal Investigator — Jewish General Hospital/McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada